CLINICAL TRIAL: NCT07380672
Title: IMpact of Mind-body Therapies (HYpnosis and Relaxation) on Anxiety in Children, Adolescents and Young Adults Who Had Been Treated in ONcology. Multicenter Study.
Acronym: HARMONY-Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23CH130; 2022-060 (Other Grant/Funding Number: INCA (French National Institute of Cancer)); ANSM (Other: 2025-A02337-42)
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Cancer Survivors; Childhood Cancer Survivors; Anxiety
Keywords: childhood cancer survivor; anxiety; depression; psychology; body mind therapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: This interventional study is divided into two studies, based on patient age, entitled HARMONY-Kids for 7-14 year olds and HARMONY-AYA for 15-25 year olds.
  The HARMONY-Kids and HARMONY-AYA studies are multicenter, prospective, randomized, open-label clinical trials comparing two treatment strategies :
  * A control group consisting of patients receiving "usual psychological care" (Group 1),
  * An experimental group consisting of patients receiving "usual psychological care + psychocorporal therapy (hypnosis or relaxation)" (Group 2).
  Centralized randomization, stratified by center and by the time between diagnosis and inclusion (≤ 18 months / > 18 months), will be performed for each of the two studies, using dedicated software. The various therapies will last six months.
  The respective populations of these two studies will be analyzed separately and will never be merged or compared with each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard psychological care (Active Comparator): Conventional follow-up. 9 sessions of standard psychological care to be completed within a maximum of 6 months (1 session every 2 weeks for 2 months, then 1 session per month for 4 months).
  Interventions: Behavioral: 9 sessions of standard psychological care
- Standard psychological care + mind-body therapy (Experimental): Standard psychological care (conventional follow-up) + psychocorporal therapy over the same period, with the patient choosing between relaxation and hypnosis
  Interventions: Behavioral: 10 mind-body therapy sessions (hypnosis or relaxation, depending on the patient's choice); Behavioral: 9 sessions of standard psychological care

INTERVENTIONS:
Behavioral: 10 mind-body therapy sessions (hypnosis or relaxation, depending on the patient's choice) — 10 sessions to be completed within a maximum of 6 months (1 session every 2 weeks for 4 months, then 1 session per month for 2 months). Sessions conducted alternately or on the same day as conventional psychotherapy sessions.
  Arms: Standard psychological care + mind-body therapy
Behavioral: 9 sessions of standard psychological care — 9 sessions of standard psychological care to be completed within a maximum of 6 months (1 session every 2 weeks for 2 months, then 1 session per month for 4 months).

SUMMARY:
In France today, it is estimated that one in 850 people aged between 20 and 45 has been cured of cancer in childhood. Some descriptive studies have established that cancer diagnosis and treatment can affect psychological health, with an increased risk of depression, post-traumatic stress, anxiety and suicidal risk. A French study published by our team in 2015 and 2020 also showed that, as adults, 40% of former pediatric cancer patients experienced symptoms of anxiety, a rate significantly higher than that of the general French population (25%).

While it is well established that it is essential to detect the onset of anxiety-depressive disorders and, if necessary, to set up conventional psychological treatment (CPT), few studies have sought to show the benefit of complementing this conventional CPT with mind-body therapies (MBT) in the post-cancer pediatric setting.

This project aims to determine the benefit of mind-body therapies (hypnosis and relaxation) as a complement to conventional psychological treatment (CPT) in the management of anxiety in children, adolescents and young adults in remission from pediatric cancer or leukemia.

ELIGIBILITY:
Inclusion Criteria:

HARMONY KIDS

* Patients aged at least 7 and under 15 at the time of inclusion, diagnosed with pediatric cancer,
* Patients considered to be in complete remission from pediatric cancer, whose intensive treatment ended at least 3 months prior to inclusion
* Patients receiving follow-up care after pediatric cancer at one of the participating centers,
* Patients with anxiety disorders (SCARED-R score ≥ 31)
* Patients affiliated with or eligible for social security,
* Patients and their parents (or legal guardians) who have received informed consent about the study and co-signed, with the investigator, a consent form to participate in the study.

HARMONY AYA

* Patients aged at least 15 and no more than 25 years old at the time of inclusion, diagnosed with pediatric cancer before the age of 18,
* Patients considered to be in complete remission from pediatric cancer, whose intensive treatment ended at least 3 months prior to inclusion,
* Patients receiving follow-up care after pediatric cancer at one of the participating centers,
* Patients with anxiety disorders (HADS-Anxiety score ≥ 8)
* Patients affiliated with or eligible for social security,
* For adult patients: patients who have received informed information about the study and have co-signed, with the investigator, a consent form to participate in the study,
* For minors: patients and their parents (or legal guardians) who have received informed consent about the study and have co-signed, with the investigator, a consent form for participation in the study.

Exclusion Criteria:

HARMONY-Kids

* Patients suffering from severe depression (CDI score > 40),
* Patients with suicidal thoughts regardless of their CDI score,
* Patients experiencing a cancer relapse,
* Refusal to participate,
* Pregnant women, women in labor, breastfeeding mothers,
* Persons deprived of their liberty, hospitalized without consent, hospitalized for purposes other than research,
* Persons subject to legal protection measures (guardianship-curatorship) or unable to express their consent HARMONY-AYA
* Patients suffering from severe depression (HADS-Depression score > 19)
* Patients with suicidal thoughts regardless of their HADS-Depression score,
* Patients with cancer relapse,
* Refusal to participate,
* Pregnant women, women in labor, breastfeeding mothers
* Persons deprived of their liberty, hospitalized without consent, hospitalized for purposes other than research
* Adults subject to legal protection measures (guardianship-curatorship) or unable to give consent.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 558 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on anxiety level in subjects aged 7 to 14 years old in remission from cancer or pediatric leukemia, compared to conventional psychological care alone. | 6 months after the first conventional psychotherapy session
  Established according to the reference scale SCARED-51 (screen for child anxiety related disorders). On this scale, each item is rated from 0 (rarely) to 2 (often), assessing the intensity of the symptom over the previous 3 months. The total score, ranging from 0 to 102 for the SCARED-R-51, is calculated by adding up the scores for all items. The higher the score, the more severe the anxiety symptoms.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on anxiety level in subjects aged 15 to 25 years old in remission from cancer or pediatric leukemia, compared to conventional psychological care alone. | 6 months after the first conventional psychotherapy session
  Established according to the Hospital Anxiety and Depression Scale (HADS). This scale comprises 14 items: 7 items relate to anxiety and 7 others to depression, allowing two separate scores to be obtained. Each response is rated from 0 to 3 on a scale that semi-quantitatively assesses the intensity of the symptom over the past week. The score for each part (anxiety/depression) is calculated by adding the values of the responses to the 7 corresponding items. Threshold scores for the two HAD subscales have been determined with the following values: 7 or less: no case, 8 to 10: doubtful case, and 11 and above: definite case.

SECONDARY OUTCOMES:
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on anxiety level in subjects aged 7 to 14 years old in remission from cancer or pediatric leukemia, compared to conventional psychological care alone. | 12 months after the first conventional psychotherapy session
  Established according to the reference scale SCARED-51 (screen for child anxiety related disorders). On this scale, each item is rated from 0 (rarely) to 2 (often), assessing the intensity of the symptom over the previous 3 months. The total score, ranging from 0 to 102 for the SCARED-R-51, is calculated by adding up the scores for all items. The higher the score, the more severe the anxiety symptoms.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on anxiety level in subjects aged 15 to 25 years old in remission from cancer or pediatric leukemia, compared to conventional psychological care alone. | 12 months after the first conventional psychotherapy session
  Established according to the Hospital Anxiety and Depression Scale (HADS). This scale comprises 14 items: 7 items relate to anxiety and 7 others to depression, allowing two separate scores to be obtained. Each response is rated from 0 to 3 on a scale that semi-quantitatively assesses the intensity of the symptom over the past week. The score for each part (anxiety/depression) is calculated by adding the values of the responses to the 7 corresponding items. Threshold scores for the two HAD subscales have been determined with the following values: 7 or less: no case, 8 to 10: doubtful case, and 11 and above: definite case.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on the level of depression in subjects aged 7 to 14 years in remission from cancer or pediatric leukemia, compared to conventional psychological care alone | 6 months then 12 months after the first conventional psychotherapy session
  Established according to the reference scale CDI (child anxiety related disorders). The CDI scale comprises 27 items, each of which is scored from 0 (absent or normal behavior for age) to 2 (severe), assessing the intensity of the symptom during the previous two weeks. The total score, ranging from 0 to 54, is calculated by adding up the scores for all items. The higher the score, the more pronounced the depressive symptoms.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on the level of depression in subjects aged 15 to 25 years in remission from cancer or pediatric leukemia, compared to conventional psychological care alone | 6 months then 12 months after the first conventional psychotherapy session
  Established according to the Hospital Anxiety and Depression Scale (HADS). This scale comprises 14 items: 7 items relate to anxiety and 7 others to depression, allowing two separate scores to be obtained. Each response is rated from 0 to 3 on a scale that semi-quantitatively assesses the intensity of the symptom over the past week. The score for each part (anxiety/depression) is calculated by adding the values of the responses to the 7 corresponding items. Threshold scores for the two HAD subscales have been determined with the following values: 7 or less: no case, 8 to 10: doubtful case, and 11 and above: definite case.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on the quality of life of subjects aged 7 to 25 in remission from pediatric cancer or leukemia, compared to conventional psychological care alone. | 6 months then 12 months after the first conventional psychotherapy session
  Established according to the Pediatric Quality of Life Inventory (PesQL). The Peds-QL measures the quality of life associated with the health status of children/adolescents in four areas: physical (8 questions), emotional (5 questions), social (5 questions), and academic (5 questions). For each question, there are 5 possible answers rated from 0 to 4 (0=never to 4=almost always) on a 5-point Likert scale or, in the version for children aged 5 to 7, 3 possible answers (0=never, 2=sometimes, and 4=almost always) on a 3-point Likert scale using smiley faces. The closer the total score, calculated as the average of all 23 questions, is to 100, the better the child/adolescent's quality of life.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on the coping strategies of subjects aged 7 to 17 in remission from pediatric cancer or leukemia, compared to conventional psychological care alone. | 6 months then 12 months after the first conventional psychotherapy session
  Established according to the reference scale KidCOPE (Coping Orientation to Problems Experienced). It is a self-administered questionnaire that has been developed in two versions, one consisting of 15 items for children aged 7 to 12, and the other consisting of 10 items for adolescents aged 13 to 18. In both cases, two dimensions are measured: frequency and effectiveness. Frequency is measured on a 4-point Likert scale. Effectiveness is measured using a 4-point Likert scale for the version for younger children (7-12 years old) and a 5-point scale for the version for older children (13-18 years old), ranging from "not helpful" to "very helpful." The results consist of a percentage of the number of subjects using each of the different coping strategies.
Evaluate the benefits of mind-body therapy as a complement to conventional psychological care on the coping strategies of subjects aged 18 to 25 in remission from pediatric cancer or leukemia, compared to conventional psychological care alone. | 6 months then 12 months after the first conventional psychotherapy session
  Established according to the reference scale BriefCOPE (Coping Orientation to Problems Experienced). This is a self-administered questionnaire consisting of 28 items, comprising 14 scales. The 14 scales of the inventory all contain two items rated from 1 to 4 (1=not at all, 2=occasionally, 3=often, and 4=always), and the score for each scale is always between 2 and 8. The results are presented as the average score for each scale of the inventory for all subjects; there is no overall score.
Determine the proportion of refusals to follow a course of treatment that includes psychological care. | through study completion, an average of 1 year
  The proportion of subjects aged 7 to 25 who refuse a course of treatment including psychological care will be determined by the number of refusals to participate in the study.
Determine the proportion of non-adherence to a care pathway that includes psychological support. | through study completion, an average of 1 year
  Non-adherence to the psychological care program proposed in this study will be determined by the termination of sessions, at the initiative of the patient or the psychologist, before reaching the minimum number of sessions required, i.e., 5 psychotherapy sessions in group 1 (arm "Usual psychological care") or 5 psychotherapy sessions combined with 5 mind-body therapy sessions in group 2 ("Usual psychological care + mind-body therapy" arm).

CONTACTS AND LOCATIONS:
Overall Officials: CLAIRE BERGER, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (7):
- France (7):
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier Universitaire Caen Normandie, Caen
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon
  - Centre Hospitalier Universitaire, Rouen
  - CENTRE HOSPITALIER UNIVERSITAIRE - site NORD, Saint-Etienne
  - CENTRE HOSPITALIER UNIVERSITAIRE - site HAUTEPIERRE, Strasbourg